CLINICAL TRIAL: NCT06001398
Title: Parent Acceptance and Commitment Therapy (PACT) for Parents of Children With Pediatric Feeding Disorder
Acronym: PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Dana Bakula, Principal Investigator, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STUDY00002540; K23MH133874 (NIH)
Record Dates: First submitted 2023-07-27; First posted 2023-08-21 (Actual); Results first posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Feeding Disorder, Chronic; Pediatric Feeding Dysfunction, Acute
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent Acceptance and Commitment Therapy (PACT) (Experimental): PACT-F is a 2-session intervention based on the Focused Acceptance and Commitment Therapy treatment literature.
  Interventions: Behavioral: Parent Acceptance and Commitment Therapy (PACT)
- Control (Active Comparator): The content of the control intervention covers a range of nutrition and healthy lifestyle topics including USDA's MyPlate.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Parent Acceptance and Commitment Therapy (PACT) — PACT is a 2-session intervention based on the Focused Acceptance and Commitment Therapy treatment literature
  Arms: Parent Acceptance and Commitment Therapy (PACT)
Behavioral: Control — The content of the control intervention covers a range of nutrition and healthy lifestyle topics including USDA's MyPlate
  Arms: Control

SUMMARY:
This is a pilot study of randomized clinical trial of Parent Acceptance and Commitment Therapy (PACT) vs. an attention-control condition (placebo) for improving the mental health of parents of children with pediatric feeding disorder.

The goal of this clinical trial is to compare two programs in parents of children with pediatric feeding disorders.

The main question[s] it aims to answer are:

* PACT will result in clinically meaningful reductions in Mental Health(MH) problems among parents of children with Pediatric Feed Disorder (PFD)
* Identify factors that impact the feasibility of PACT delivery

  * Participants will asked to participate in one of two programs focused on parents of children with pediatric feeding disorders.
  * The participants will also be asked to complete a battery of questionnaires at four timepoints during the study.
  * The parents will be asked to video record a meal time twice during study.

If there is a comparison group: Researchers will compare the PACT group with a control group to see if PACT will result in clinically meaningful change in parent stress and anxiety, and parent use of positive mealtime behaviors.

DETAILED DESCRIPTION:
The goal of this study is to advance the science of a brief parent mental health intervention for parents of children with pediatric feeding disorder using Parent Acceptance and Commitment Therapy (PACT-F). The ultimate goal of this research is to improve parent mental health and child health and feeding outcomes through a parent-focused behavioral intervention.

PACT-F is a 2-session acceptance and commitment therapy (ACT) intervention guided by Brown and Whittingham's ACT intervention for parents of children with neurodevelopmental conditions. Intervention content is based on principles of ACT, an evidence-based treatment for adult mental health problems. The intervention content is therefore broadly applicable to all parents but was specifically tailored for the needs of parents of children with neurodevelopmental conditions. In study phase 1 of this award, the investigators adapted parent ACT for parents of children with pediatric feeding disorder (PACT-F) with consultation from 2 parents of children with pediatric feeding disorder and 2 experts in parent ACT. The investigators now have a complete treatment package that has been tailored for parents of children with pediatric feeding disorder and is ready to be piloted.

Thus, in this study the investigators will conduct a feasibility and proof-of-concept pilot of a 2-session parent-focused ACT intervention tailored to meet the needs of parents of children with pediatric feeding disorder (PACT-F). The goal of this pilot is to determine factors that impact the success of recruitment, retention, assessment, and treatment delivery for the PACT-F clinical trial and to test the intervention's proof of concept (i.e., does it show a clinically meaningful signal of change in parent mental health). This study will be conducted at a single site (Children's Mercy Hospital). The investigators will pilot the clinical trial procedures and monitor feasibility success, and factors that may impact feasibility success. Participants who meet inclusion criteria will be randomized to either PACT-F or an attention control (control) condition. Participants will be blind to treatment condition (single blind study). The aim of the feasibility analyses is to evaluate factors critical to success, rather than evaluating whether the intervention is "feasible or not feasible". The aim of the proof-of-concept analyses is to determine if this intervention has promise and warrants a larger efficacy trial.

Parents randomized to PACT-F will complete two 90-minute PACT-F sessions individually with a study interventionist, 2 weeks apart. Parents randomized to the control group will complete two 90-minute sessions individually with a study interventionist, 2-weeks apart (focused on nutrition education). The control intervention will be parallel to the ACT intervention in all ways, including interactive components and the face-to-face time with health professionals (interventionists). The control condition intervention has already been developed by Dr. Davis's research team and covers a range of nutrition and healthy lifestyle topics including the United States Department of Agriculture's (USDA) MyPlate. An attention control condition was selected to mimic the interpersonal benefits that may come from meeting individually with a caring professional. The control condition intervention content (healthy lifestyles) was specifically chosen as it most closely reflects the types of information that parents would learn from healthcare professionals about the type of nutrition that their child needs. However, this type of intervention should not impact parent mental health.

Interventionists for both conditions will be individuals with at least master's degree training in mental health or a related field. The interventions will take via tele-video conferencing to allow participants to participate from home without needing transportation to and from the hospital. Both arms of the intervention will be manualized and interventionists in both arms will be trained using didactics and role playing with the Principle Investigator(PI). Intervention fidelity will be monitored by audio/video recording all sessions. The PI (Dr. Bakula) will review recordings each week and conduct separate 1-hour weekly supervision of study interventionists for each arm of the study (PACT-F & control).

Strategies will be used to promote fidelity in line with recommendations from the NIH Behavior Change Consortium. A fidelity checklist will be developed in line with adaptations to the intervention and will be piloted with study interventionists. The fidelity checklist will be refined during research team meetings. The fidelity checklist will be reviewed by the PI during supervision.

Hypothesis testing: The investigators will test the hypothesis that PACT-F results in clinically meaningful change using the Reliable Change Index (RCI; success defined as RCI > 1.96). The investigators anticipate that these procedures will be feasible, with feasibility success defined as recruitment rate above 60%, and retention, assessment completion, and intervention completion rate above 80%. Mixed methods data collection will identify factors that impact 1) recruitment rate (qualitative interviews, % meeting inclusion criteria, # of contact attempts), 2) retention rates (qualitative interviews, baseline characteristics; treatment group), 3) assessment completion rate (qualitative interviews, measure type), and 4) treatment completion rate (qualitative interviews, scheduling, treatment location).

The proposed study is an important first step towards developing an evidence-based treatment that can be used with parents of children with pediatric feeding disorder. This intervention has the potential to improve parent mental health, as well as child health, and therefore has the potential to have broad public health impact.

ELIGIBILITY:
Inclusion Criteria:

* 1) Must be a parent aged 18+ (primary caregiver) of 2-6-year-old child with PFD
* 2) Child must be receiving outpatient PFD treatment at Children's Mercy Hospital (CMH)
* 3) The parent must have a clinically significant elevation on at least one measure of parent MH (using established clinical cutoffs). Parents will be included regardless of whether the child has a new diagnosis or established diagnoses

Exclusion Criteria:

* 1) Parent has significant cognitive impairments
* 2) Parent does not speak English
* Parent unable to obtain high speed internet at home

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana Bakula, PhD, Principal Investigator — Children's Mercy Hosptial
Locations (1):
- Children's Mercy Hospitals and Clinics, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Parent Acceptance and Commitment Therapy (PACT) | Control
Started | 20 | 10
Completed | 14 | 6
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parent Acceptance and Commitment Therapy (PACT) | Control | Total
Number analyzed (Participants) | 14 | 6 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (8.39) | 31 (6.66) | 34 (7.96)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 0 | 2
  White | 12 | 5 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 13 | 6 | 19
  Unknown or Not Reported | 0 | 0 | 0
PHQ9 [Mean (Standard Deviation); unit: Rating Scale] — PATIENT HEALTH QUESTIONNAIRE-9. The scale has a possible range of 0 to 27, with higher scores indicating worse depression.
  Rating Scale | 6.57 (4.48) | 7.33 (3.56) | 6.80 (4.15)
GAD7 [Mean (Standard Deviation); unit: Rating Scale] — Generalized Anxiety Disorder 7-item (GAD-7). The scale has a possible range of 0 to 21, with higher scores indicating worse anxiety.
  Rating Scale | 8.64 (4.85) | 8.83 (3.66) | 8.70 (4.43)
PSS [Mean (Standard Deviation); unit: Rating Scale] — Perceived Stress Scale. The scale has a possible range of 0 to 40, with higher scores indicating worse stress.
  Rating Scale | 21.21 (5.24) | 18.83 (4.71) | 20.50 (5.08)
IESR [Median (Standard Deviation); unit: Rating Scale] — IMPACT OF EVENTS SCALE-Revised (IES-R). The scale has a possible range of 0 to 88, with higher scores indicating worse posttraumatic stress symptoms.
  Rating Scale | 23.93 (19.99) | 22.17 (18.43) | 23.40 (19.07)
BPFAS [Mean (Standard Deviation); unit: Rating Scale] — Behavioral Pediatrics Feeding Assessment Scale (Total Frequency Score). The scale has a possible range of 35 to 175, with higher scores indicating worse feeding problems.
  Rating Scale | 91 (11.49) | 96.14 (14.10) | 92.5 (12.22)

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a 9-item self-report measure of depressive symptoms. We used the Reliable Change Index to determine if within-person change was obtained for each participant in the treatment group. Within person change was The Reliable Change Index (RCI) is calculated using a formula that takes into account the pre-test score, post-test score, standard deviation of the test and test-retest reliability coefficient. If the computed within-person value exceeds +/- 1.96 it is considered a significant change. For this study, we then counted the number of participants who had significant improvements in this outcome variable compared to those who did not.
Time Frame: Measured 2-week post-intervention
Population: This outcome measure is only assessed in the active treatment group as it was pre-specified that this data is only pertinent to the active treatment group being assessed. This was a proof of concept study and the control group was only completed for feasibility/acceptability evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Acceptance and Commitment Therapy (PACT) | Control
Number analyzed (Participants) | 14 | 0
Participants
  Significant Reliable Change Index Score | 2 | 0
  Non-Significant Reliable Change Index Score | 12 | 0

2. Primary Outcome: General Anxiety Disorder Screener (GAD-7)
Description: The GAD-7 is a 7-item self-report measure of anxious symptoms. We used the Reliable Change Index to determine if within-person change was obtained for each participant in the treatment group. Within person change was The Reliable Change Index (RCI) is calculated using a formula that takes into account the pre-test score, post-test score, standard deviation of the test and test-retest reliability coefficient. If the computed within-person value exceeds +/- 1.96 it is considered a significant change. For this study, we then counted the number of participants who had significant improvements in this outcome variable compared to those who did not.
Time Frame: Measured 2-week post-intervention
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Acceptance and Commitment Therapy (PACT) | Control
Number analyzed (Participants) | 14 | 0
Participants
  Significant Reliable Change Index Score | 4 | 0
  Non-Significant Reliable Change Index Score | 10 | 0

3. Primary Outcome: Impact of Event Scale - Revised (IES-R)
Description: The IES-R is a 22-item self-report measure of posttraumatic stress symptoms. We used the Reliable Change Index to determine if within-person change was obtained for each participant in the treatment group. Within person change was The Reliable Change Index (RCI) is calculated using a formula that takes into account the pre-test score, post-test score, standard deviation of the test and test-retest reliability coefficient. If the computed within-person value exceeds +/- 1.96 it is considered a significant change. For this study, we then counted the number of participants who had significant improvements in this outcome variable compared to those who did not.
Time Frame: Measured 2-week post-intervention
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Acceptance and Commitment Therapy (PACT) | Control
Number analyzed (Participants) | 14 | 0
Participants
  Significant Reliable Change Index Score | 2 | 0
  Non-Significant Reliable Change Index Score | 12 | 0

4. Primary Outcome: Perceived Stress Scale (PSS)
Description: The PSS is a 10-item self-report measure of perceived stress. We used the Reliable Change Index to determine if within-person change was obtained for each participant in the treatment group. Within person change was The Reliable Change Index (RCI) is calculated using a formula that takes into account the pre-test score, post-test score, standard deviation of the test and test-retest reliability coefficient. If the computed within-person value exceeds +/- 1.96 it is considered a significant change. For this study, we then counted the number of participants who had significant improvements in this outcome variable compared to those who did not.
Time Frame: Measured 2-week post-intervention
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Acceptance and Commitment Therapy (PACT) | Control
Number analyzed (Participants) | 14 | 0
Participants
  Significant Reliable Change Index Score | 3 | 0
  Non-Significant Reliable Change Index Score | 11 | 0

5. Primary Outcome: Behavioral Pediatrics Feeding Assessment Scale (BPFAS)
Description: Behavioral Pediatrics Feeding Assessment Scale (Total Frequency Score). The scale has a possible range of 35 to 175, with higher scores indicating worse feeding problems. The BPFAS is a 35-item parent-proxy report of child mealtime and feeding behavior. This was not evaluated using the RCI and instead was only a metric evaluated for pre-post scores in the intervention group as it was an exploratory assessment.
Time Frame: Measured 2-week post-intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Rating Scale
Arm/Group | Parent Acceptance and Commitment Therapy (PACT) | Control
Number analyzed (Participants) | 14 | 0
Rating Scale | 88.69 (12.53) |

6. Primary Outcome: Retention Rate
Description: This is a measure of the % of participants who were able to be retained from baseline through to the end of the study (3 month follow up). This was assessed as a component of feasibility.
Time Frame: 3-month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Acceptance and Commitment Therapy (PACT) | Control
Number analyzed (Participants) | 20 | 10
Participants | 14 | 6

7. Primary Outcome: Intervention Completion Rate
Description: This is a measure of the % of participants who started the intervention, and then successfully completed all sessions. This was assessed as a component of feasibility.
Time Frame: Intervention Completion (2 week follow up)
Population: For participants who began the first session of the intervention (n=14 in the PACT arm, n=6 in the Control arm), this is the number of participants who subsequently completed both intervention sessions in full.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Acceptance and Commitment Therapy (PACT) | Control
Number analyzed (Participants) | 14 | 6
Participants | 14 | 6

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from enrollment to study completion at 3 month follow up or time of withdrawal from the study.
Description: Adverse events were defined in line with clinicaltrials.gov and NIH definitions.
Arm/Group | Parent Acceptance and Commitment Therapy (PACT) | Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 0/20 | 0/10

LIMITATIONS AND CAVEATS:
The findings of this study should be interpreted with caution as this was a pilot study focused on feasibility, acceptability, and proof-of-concept in a small sample of families. Further research is needed to assess efficacy of this intervention through a large, appropriately powered randomized clinical trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Study protocol and Statistical Analysis Plan v. 2 (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT06001398/Prot_SAP_000.pdf